CLINICAL TRIAL: NCT04391296
Title: Prospective Randomized Control Study About the Effect of Postmastectomy Radiation Therapy on Capsular Contracture in Patients With Prepectoral or Subpectoral Implant-based Breast Reconstruction: PREPER Trial
Brief Title: Capsular Contracture After PMRT Using Prepectoral Versus Subpectoral Implant-based Breast Reconstruction: PREPER Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0837-002
Record Dates: First submitted 2020-05-03; First posted 2020-05-18 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast implants
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I (Prepectoral) (Experimental): Immediate acellular dermal matrix-assisted implant-based breast reconstruction with prepectoral implant placement.
  Interventions: Procedure: Arm I (Prepectoral), Arm II (Subpectoral)
- II (Subpectoral) (Active Comparator): Immediate acellular dermal matrix-assisted implant-based breast reconstruction with subpectoral implant placement.
  Interventions: Procedure: Arm I (Prepectoral), Arm II (Subpectoral)

INTERVENTIONS:
Procedure: Arm I (Prepectoral), Arm II (Subpectoral) — Arm I (Prepectoral)De-epithelialized skin flaps are made from the inferior pole of breast skin and soft tissue. The implant pocket is shaped by fixing a sufficiently large amount of ADM to the medial surface of the mastectomy pocket, the upper edge of the pectoralis major muscle and the de-epithelial skin flap. The implant is located in the prepectoral mastectomy pocket and the ADM anchored to the chest wall, serratus fascia, and de-epithelial skin flaps. The pectoralis major muscle is located in the anatomical location behind the ADM.
  Arm II (Subpectoral)The pectoralis major muscle is dissected from the thorax to create sufficient space for the implant to be placed behind the pectoralis major muscle. Implant pockets are made by suturing the lower part of the elevated pectoralis major muscle to the top of the de-epithelial skin flap and the ADM patch to the skin flap, the pectoralis major muscle, and the lateral thoracic fascia.

SUMMARY:
The purpose of this study is to prospectively compare and analyze the incidence of complications in patients undergoing postmastectomy radiation therapy after breast reconstruction with subpectoral and prepectoral placement of implant. Investigators hypothesized that immediate acellular dermal matrix-assisted implant-based breast reconstruction with prepectoral implant placement would result in lower risk of capsular contracture after postmastectomy radiation therapy(PMRT) compared with acellular dermal matrix(ADM)-assisted implant-based breast reconstruction with subpectoral implant placement.

DETAILED DESCRIPTION:
OUTLINE: This is a single center randomized clinical trial. Participant recruitment and enrollment will occur at Gangnam Severance Hospital Breast Cancer Center for 4 years, followed by one year of follow up data collection and analysis.

Arm I (Prepectoral): immediate ADM-assisted implant-based breast reconstruction with prepectoral implant placement.

Arm II (Subpectoral): immediate ADM-assisted implant-based breast reconstruction with subpectoral implant placement.

This clinical study is aimed at patients who have been diagnosed with breast cancer and who have undergone a total mastectomy for the therapeutic indication, and who are planning to undergo implant based reconstruction and postmastectomy radiotherapy.

It will be carried out prospectively in a single institution, and the study will be divided into two groups, subpectoral implant and prepectoral implant, according to the reconstruction method.

A total of 96 patients or 48 patients per arm will be recruited. Randomization will be accomplished using randomly permuted blocks, and randomization will be stratified on the basis of reconstruction method. (tissue expander insertion or direct-to-implant)

After completion of study treatment, patients are followed for 1 year for observation of capsular contracture and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 19 years old
2. Histologically confirmed diagnosis of unilateral breast cancer
3. Mastectomy (nipple or skin sparing mastectomy) candidate for therapeutic indication
4. Patient undergoing immediate implant based breast reconstruction

Exclusion Criteria:

1. Underlying medical condition: for example, (AST or ALT >100U/L, inadequate renal function; eGFR < 30ml/min, congestive heart failure; New York Heart Association III-IV)
2. Prior history of radiotherapy on the affected side of breast or chest wall before mastectomy
3. History of a known additional malignancy Note: Participants with melanoma of skin, low grade thyroid cancer are not excluded.
4. Not able to provide informed consent (Illiterate, foreigners, etc.)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of capsular contracture (grade 3 or higher) (%) by Baker's scale | 6 months after the completion of PMRT
  To compare the frequency of grade 3 or higher contracture development analyzed by using Baker's scale at 6 months after the completion of PMRT.
Rate of capsular contracture (grade 3 or higher) (%) by 2D shear elastography | 6 months after the completion of PMRT
  To compare the frequency of grade 3 or higher contracture development analyzed by using 2D shear-wave elastography at 6 months after the completion of PMRT.

SECONDARY OUTCOMES:
Patient reported outcome | 1 year after the completion of PMRT
  1) To compare the patient reported outcome (PRO) using Breast Q questionnaire (Reconstruction module, each domain has the scale ranges from 0 to 100, higher the better patient reported outcome)
Rate of capsular contracture (grade 3 or higher) (%) in long term follow up | 1 year after the completion of PMRT
  1) To compare the rate of Grade 3 or higher capsular contracture at 1 year after the end of PMRT